CLINICAL TRIAL: NCT01559168
Title: Clinical Evaluation of the Uphold Mesh for the Surgical Treatment of Uterine-predominant Prolapse: a Prospective, Multicenter Trial
Brief Title: Uphold Mesh for the Surgical Treatment of Uterine-predominant Prolapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LOCAL/2011/RdeT-04; 2011-A01705-36 (Other: ANSM)
Record Dates: First submitted 2012-03-19; First posted 2012-03-21 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2017-01

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prolapse patients recieving UpHold LITE (Experimental): Non-pregnant female patients >= 50 years who are not considering future pregnancies, who are diagnosed with uterine or vault prolapse with ICS POP-Q score of stage 2 or greater, who are receiving the UpholdTM LITE mesh kit and who agree to be in the study.
  Interventions: Device: UpholdTM LITE placement

INTERVENTIONS:
Device: UpholdTM LITE placement — Uphold TM LITE mesh is used for the surgical correction of pelvic organ prolapse.

SUMMARY:
The primary objective of this study is to evaluate the efficacy of the UpholdTM LITE mesh over a 12 month follow up period, using a composite outcome including a good anatomical correction for both anterior and apical compartments (stage 0 or 1), no prolapse (bulge) symptoms (answer "no" at question 3 of the PFDI-20) and no reintervention for recurrent prolapse of the anterior or apical compartment.

DETAILED DESCRIPTION:
Secondary objectives include the evaluation of the following:

* Change from baseline of POP-Q scoring at 6 weeks, 6 months and 12 months post procedure, including evolution of treated or non-treated posterior compartments.
* The proportion of patients with anatomical prolapse (C/D), but who are asymptomatic.
* Change from baseline of mean quality-of-life scores.
* Evaluation of mesh properties from procedure date through study period.
* Peri-operative and post-treatment pain score assessment comparing the various anesthesia regimes used (Visual Analog Scale).
* Assessment of patient subjective outcomes for overall treatment effects and satisfaction.
* Objective evaluation of mesh shrinkage by standardized ultrasound measurements.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is available for 12 months of follow-up
* Patients with symptoms and altered quality of life in relation to uterine or post-hysterectomy vault prolapse
* Patients who are receiving the UpholdTM LITE mesh Kit
* Female patients >= years who have no desire of future pregnancy
* Diagnosed with pelvic organ prolapse and >= ICS POP-Q Stage 2 Symptomatic Prolapse apical compartment (uterine or vault), associated with ICS POP-Q Stage 2 or 3 Symptomatic Prolapse anterior compartment (point Ba >= -1
* Patients willing to complete quality of life questionnaire at baseline (pre-procedure) and at 6 weeks, 6 and 12 months post-procedure

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant, parturient, or breastfeeding
* Patients who are not receiving the UpHoldTM LITE mesh Kit
* Patients < 50 years
* Patients qho, according to the clinical judgment of the investigator, are not suitable for this study
* Patients who are considering future pregnancies
* Patients whose pelvic organ prolapse is a <= 1 ICS Stage
* Patients requiring Posterior Graft procedure
* Patients with known or suspected hypersensitivity to polypropylene
* Patients with any pathology which ould compromise implant placement
* Patients with any pathology which ould compromise implant placement as mentioned in the device instruction manual
* Patients with any pathology that would limit blood supply and compromise healing
* Patients with blood coagulation disorder (associated current level coagulation)
* Patients with autoimmune connective tissue disease
* Patients with upper urinary tract obstruction and renal insufficiency
* Patients with local or systemic infection

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2012-10; Primary Completion 2016-10-12 (Actual); Study Completion 2016-10-12 (Actual)

PRIMARY OUTCOMES:
Apical anatomical success | 12 months
  Presence/absence: anatomical success as concerns apical (uterine) support, defined as point C <= stage 1 per POP-Q scoreing (ICS)
Anterior vaginal wall anatomical success | 12 months
  Presence/absence: anatomical success on anterior vaginal wall support, defined as point Ba < = stage 1 per POP-Q scoring (ICS)
Change from baseline in PFDI-20 scores | baseline to 12 lines

SECONDARY OUTCOMES:
Anterior vaginal wall anatomical success | 6 months
  Presence/absence: anatomical success on anterior vaginal wall support, defined as point Ba < = stage 1 per POP-Q scoring (ICS)
Apical anatomical success | 6 weeks
  Presence/absence: anatomical success as concerns apical (uterine) support, defined as point C <= stage 1 per POP-Q scoreing (ICS)
Apical anatomical success | 6 months
  Presence/absence: anatomical success as concerns apical (uterine) support, defined as point C <= stage 1 per POP-Q scoreing (ICS)
Anterior vaginal wall anatomical success | 6 weeks
  Presence/absence: anatomical success on anterior vaginal wall support, defined as point Ba < = stage 1 per POP-Q scoring (ICS)
Change from baseline in PFDI-20 scores | baseline to 6 weeks
Change from baseline in PFDI-20 scores | baseline to 6 months
Change from baseline in PFIQ-7 scores | baseline to 6 weeks
Change from baseline in PFIQ-7 scores | baseline to 6 months
Change from baseline in PFIQ-7 scores | baseline to 12 months
Change from baseline in PISQ-12 scores | baseline to 6 months
Change from baseline in PISQ-12 scores | baseline to 12 months
length of hospital stay (days) | 6 weeks
Number of days necessary for return to normal activities | 6 weeks
Visual analog scale for post-operative pain | Day 1
  score ranging from 0.0 to 10.0
Visual analog scale for post-operative pain | 6 weeks
  score ranging from 0.0 to 10.0
Visual analog scale for post-operative pain | 6 months
  score ranging from 0.0 to 10.0
Visual analog scale for post-operative pain | 12 months
  score ranging from 0.0 to 10.0
Mesh related morbidity | Day 1
  Presence/absence of mesh related morbidity (infection, erosion, pain, dyspareunia)
Mesh related morbidity | 6 weeks
  Presence/absence of mesh related morbidity (infection, erosion, pain, dyspareunia)
Mesh related morbidity | 6 months
  Presence/absence of mesh related morbidity (infection, erosion, pain, dyspareunia)
Mesh related morbidity | 12 months
  Presence/absence of mesh related morbidity (infection, erosion, pain, dyspareunia)
Mesh contraction (cm) | 6 weeks
  Mesh contraction as determined by ultrasound measurement (cm)
Mesh contraction (cm) | 6 months
  Mesh contraction as determined by ultrasound measurement (cm)
Mesh contraction (cm) | 12 months
  Mesh contraction as determined by ultrasound measurement (cm)
Patient satisfaction (PGI index) score | 6 weeks
Patient satisfaction (PGI index) score | 6 months
Patient satisfaction (PGI index) score | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Renaud de Tayrac, MD PhD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (13):
- France (13):
  - CH Camille Guérin, Châtellerault
  - CHU de Clermont Ferrand - Hôpital Estaing, Clermont-Ferrand
  - CH de Dunkerque, Dunkirk
  - CH de Gonesse, Gonesse
  - CHRU de Lille - Hôpital Jeanne de Flandre, Lille
  - CHRU de Lyon - Hôpital de la Croix Rousse, Lyon
  - APHM - Hôpital de la Conception, Marseille
  - Clinique Beau Soleil, Montpellier
  - CHU de Montpellier - Hôpital Lapeyronie, Montpellier
  - CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes
  - CH Louis Giorgi, Orange
  - CHU de Poitiers, Poitiers
  - Hôpital Foch, Suresnes

REFERENCES:
- [Result] Allegre L, Debodinance P, Demattei C, Fabbro Peray P, Cayrac M, Fritel X, Courtieu C, Fatton B, de Tayrac R. Clinical evaluation of the Uphold LITE mesh for the surgical treatment of anterior and apical prolapse: A prospective, multicentre trial. Neurourol Urodyn. 2019 Nov;38(8):2242-2249. doi: 10.1002/nau.24125. Epub 2019 Jul 29. PMID 31359498